CLINICAL TRIAL: NCT06239558
Title: Barriers and Enablers to Cardiac Rehabilitation Uptake, Adherence and Completion Experienced by Service Users With South Asian Heritage
Brief Title: Cardiac Rehabilitation Participation and South Asian Service Users
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: Wellcome Trust (Other); University Hospitals, Leicester (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0960
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Rehabilitation; South Asian Service Users

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- South Asian Service Users: Service users who identify themselves as South Asian will be invited to participant in a semi-structured interview and/or a focus group. The interview will be used to identify lived experiences of the barriers and enablers to cardiac rehabilitation, relating to uptake, adherence or completion. The focus group will be used to collaboratively generate adaptations to CR services which could be implemented to overcome the barriers, and enhance the enablers, identified during the interviews.
  Interventions: Other: Qualitative exploration
- Cardiac Rehabilitation Healthcare Professionals: The rehabilitation healthcare professionals will be invited to participant in a semi-structured interview and/or a focus group. The interviews will be used to explore their the perceptions of barriers and enablers and knowledge around the cultural requirements of South Asian service users.
  Interventions: Other: Qualitative exploration
- Key stakeholders: Key stakeholders relating to cardiac rehabilitation, University Hospitals of Leicester (UHL) NHS Trust, and/or South Asian communities will be invited to participate in the focus group, helping to generate adaptations to CR services.
  Interventions: Other: Qualitative exploration

INTERVENTIONS:
Other: Qualitative exploration — Semi-structured Interviews and focus group

SUMMARY:
The goal of this qualitative study is to learn about the barriers and enablers to cardiac rehabilitation, experience by South Asian service users based in the UK who have experienced an acute cardiac event and been referred for CR. This may allow NHS programmes to make adaptations to their services to enhance uptake, adherence and completion for this ethnic population. The main questions it aims to answer are:

* What are the barriers and enablers to uptake, adherence or completion of CR experienced by service users with South Asian heritage?
* What adaptations to the CR service could be implemented to overcome identified barriers, enhance enablers and result in increased uptake, adherence or completion to CR?

Participants will be invited to participate in a semi-structured interview and/or a focus group to explore lived experiences that can answer the research questions.

DETAILED DESCRIPTION:
This study aims to explore contemporary barriers and enablers to uptake, adherence or completion of cardiac rehabilitation experienced by service users with South Asian heritage, and develop culturally relevant programme adaptations to overcome the identified barriers. Cardiac rehabilitation (CR) a highly evidenced exercise-based intervention offered to eligible patients who have experienced a cardiac event however South Asian service users are less likely to uptake, adhere to or complete CR. This may be because cultural acceptability of CR components (assessment, exercise and education sessions) are not fully considered or tailored for this ethnic population. This study will explore what barriers and enablers are experienced by South Asian service users, with a focus on cultural and psychosocial factors, and develop culturally relevant programme adaptations to increase uptake, adherence and completion. The study will also explore healthcare professionals (HCPs) perceptions of barriers and enablers to CR experienced by service users with South Asian heritage. Participants will include adult (≥ 18 years) service users who have a South Asian heritage and have been referred to University Hospitals of Leicester CR after a cardiac event. Participants will also include healthcare professions and key stakeholders involved in CR and health inequalities. Participants will be invited to a community-based interview (1 hour) and/or a workshop (3 hours) to provide their experiences of barriers and enablers to CR and help develop culturally appropriate service adaptations to overcome these barriers and enhance enablers, resulting increased uptake, adherence or completion of CR. The study is funded by the Wellcome Trust as part of the Leicestershire Health Inequalities Improvement Programme as the University of Leicester.

ELIGIBILITY:
Inclusion Criteria:

Service Users

* Adult aged ≥18 years
* Has capacity to give consent
* Been referred to UHL NHS Trust cardiac rehabilitation service
* Has experienced an acute cardiac event which is eligible for CR provided by UHL CR service
* Identifies their ethnicity as South Asian i.e. ancestral origins in India, Pakistan, Bangladesh, Afghanistan, Bhutan, Maldives, Nepal and Sri Lanka (Indian sub-continent).
* Workshop only: be able to communicate in spoken English

CR Healthcare Professionals

* Adult aged ≥18 years
* Has capacity to give consent
* HCP involved in delivering direct patient care, who works within UHL NHS Trust CR service

Key Stakeholders

* Adult aged ≥18 years
* Has capacity to give consent
* Individuals who have a direct involvement with South Asian communities, tackling health inequalities, NHS commissioning or service development, or CR policy/guideline development

Exclusion Criteria:

Service Users

* Child aged <18 years
* Unable to give consent
* Have not been referred to UHL NHS Trust CR services
* Been referred to CR due to heart failure and will conduct CR within a community-provided breathlessness pathway
* Does not self-identify as South Asian
* Workshop only: unable to speak or understand spoken English

CR Healthcare Professionals

* Child aged <18 years
* Unable to give consent
* Not a CR team member involved in delivering direct patient care, who works within UHL NHS Trust CR service

Key Stakeholders

* Child aged <18 years
* Unable to give consent
* Not an individual who have a direct influence on South Asian communities, tackling health inequalities, NHS commissioning or service development, or CR policy/guideline development
* Unable to attend workshop in person

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * adults referred to cardiac rehabilitation with South Asian heritage
  * cardiac rehabilitation (CR) healthcare professionals working at University of Leicester Hospitals CR service
  * key stakeholders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Identification of contemporary barriers and enablers to cardiac rehabilitation | 90 minute interviews
  Barriers and enablers to cardiac rehabilitation experienced by South Asian service users
Cardiac Rehabilitation Programme Adaptations | 3 hour interactive focus group
  Adaptations to the service which could be implemented to overcome identified barriers, enhance enablers and result in increased uptake, adherence or completion.

SECONDARY OUTCOMES:
Healthcare professionals perceptions of barriers and enablers | 90 minute interviews
  Healthcare professionals perceptions of barriers and enablers experienced by South Asian service users which may influence uptake, adherence to and completion of cardiac rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Sally J Singh, PhD, Principal Investigator — University of Leicester
Locations (1):
- Glenfield General Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No